CLINICAL TRIAL: NCT00049283
Title: A Phase I Study of the Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor, OSI-774, in Combination With Docetaxel and Radiation in Locally Advanced Squamous Cell Cancer of the Head and Neck
Brief Title: Erlotinib, Docetaxel, and Radiation Therapy in Treating Patients With Locally Advanced Head and Neck Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03113; CWRU 1301; U01CA099168 (NIH); U01CA062502 (NIH)
Record Dates: First submitted 2002-11-12; First posted 2003-01-27 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2013-01

CONDITIONS: Metastatic Squamous Neck Cancer With Occult Primary Squamous Cell Carcinoma; Stage III Squamous Cell Carcinoma of the Hypopharynx; Stage III Squamous Cell Carcinoma of the Larynx; Stage III Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage III Squamous Cell Carcinoma of the Nasopharynx; Stage III Squamous Cell Carcinoma of the Oropharynx; Stage III Verrucous Carcinoma of the Larynx; Stage III Verrucous Carcinoma of the Oral Cavity; Stage IV Squamous Cell Carcinoma of the Hypopharynx; Stage IV Squamous Cell Carcinoma of the Nasopharynx; Stage IVA Squamous Cell Carcinoma of the Larynx; Stage IVA Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IVA Squamous Cell Carcinoma of the Oropharynx; Stage IVA Verrucous Carcinoma of the Larynx; Stage IVA Verrucous Carcinoma of the Oral Cavity; Stage IVB Squamous Cell Carcinoma of the Larynx; Stage IVB Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IVB Squamous Cell Carcinoma of the Oropharynx; Stage IVB Verrucous Carcinoma of the Larynx; Stage IVB Verrucous Carcinoma of the Oral Cavity; Stage IVC Squamous Cell Carcinoma of the Larynx; Stage IVC Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IVC Squamous Cell Carcinoma of the Oropharynx; Stage IVC Verrucous Carcinoma of the Larynx; Stage IVC Verrucous Carcinoma of the Oral Cavity; Tongue Cancer; Untreated Metastatic Squamous Neck Cancer With Occult Primary
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Tongue Neoplasms | interventions — Erlotinib Hydrochloride; Docetaxel; Radiotherapy; Radiation

ARMS (1):
- Treatment (erlotinib hydrochloride, docetaxel, and radiation) (Experimental): Patients receive oral erlotinib alone daily on weeks 1 and 2. Patients then receive oral erlotinib daily beginning on day 1 and docetaxel IV over 1 hour on day 3 of weeks 3-9. Patients also undergo radiotherapy once daily 5 days a week on weeks 3-9. Patients continue erlotinib for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients who had N2 or greater cervical lymph node involvement at baseline or have residual neck adenopathy after chemoradiotherapy undergo neck dissection 6-8 weeks after completion of chemoradiotherapy. Erlotinib is held for 1 week before planned surgery and until healing is complete.
  Interventions: Drug: erlotinib hydrochloride; Drug: docetaxel; Radiation: radiation therapy; Procedure: therapeutic conventional surgery; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: erlotinib hydrochloride — Given orally
  Other Names: CP-358,774; erlotinib; OSI-774
Drug: docetaxel — Given IV
  Other Names: RP 56976; Taxotere; TXT
Radiation: radiation therapy — Undergo radiotherapy
  Other Names: irradiation; radiotherapy; therapy, radiation
Procedure: therapeutic conventional surgery — Undergo neck dissection
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Erlotinib may stop the growth of tumor cells by blocking the enzymes necessary for tumor cell growth. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining erlotinib with docetaxel may make the tumor cells more sensitive to radiation therapy and may kill more tumor cells. Phase I trial to study the maximum tolerated dose (MTD) of combining erlotinib with docetaxel and radiation therapy in treating patients who have locally advanced head and neck cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine MTD and toxicity of combination of EGFR inhibitor (OSI-774), docetaxel, and radiation.

II. Pharmacokinetic profile of OSI-774 alone and in combination with docetaxel.

SECONDARY OBJECTIVES:

I. Determine the overall and complete response rate of this combination.

II. Determine overall, disease free, and progression free survival of this combination.

* EGFR expression and phosphorylation status
* Serum markers of angiogenic activity VEGF, sVEGFR-2, sKIT, ICAM, PDGF
* Fluorescence in situ hybridization (FISH) for EGFR, ERBB2, PDGFR-β for gene amplification
* DNA-sequencing of EGFR and ERBB2 genes from DNA extracted from pretreatment biopsy material for mutation screening
* Gene expression profiling on pre-treatment biopsy material to identify predictors of response to treatment
* Apoptosis (TUNEL assay)
* Ki67 (nuclear proliferation antigen).

OUTLINE: This is a dose-escalation study of erlotinib and docetaxel.

Patients receive oral erlotinib alone daily on weeks 1 and 2. Patients then receive oral erlotinib daily beginning on day 1 and docetaxel IV over 1 hour on day 3 of weeks 3-9. Patients also undergo radiotherapy once daily 5 days a week on weeks 3-9. Patients continue erlotinib for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients who had N2 or greater cervical lymph node involvement at baseline or have residual neck adenopathy after chemoradiotherapy undergo neck dissection 6-8 weeks after completion of chemoradiotherapy. Erlotinib is held for 1 week before planned surgery and until healing is complete.

Cohorts of 3-6 patients receive escalating doses of erlotinib and docetaxel until the MTD is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed every 16 weeks for 1 year after completion of erlotinib, every 24 weeks for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: Approximately 30 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed locally advanced (stage III or IV) squamous cell carcinoma of the head and neck without distant metastatic disease
* No prior chemotherapy, radiation therapy, or investigational anti-tumor drug
* Measurable disease within 4 weeks prior to registration according to the recommended RECIST response criteria
* ECOG performance status =< 2 (Karnofsky >= 60%)
* Life expectancy of greater than 12 weeks
* Absolute neutrophil count >= 1,500/ul
* Platelets >= 100,000/ul
* Hemoglobin >= 10 mg/dL
* Total bilirubin within normal institutional limits
* AST(SGOT)/ALT(SGPT) =< 5 x ULN when alkaline phosphatase is =< ULN
* Alkaline phosphatase =< 5 x ULN when AST or ALT =< ULN
* Prothrombin time within normal institutional limits
* Creatinine within normal institutional limits or creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* No clinically significant heart disease (including NYHA class III or IV heart disease, significant arrhythmias requiring medication, symptomatic coronary artery disease, myocardial infarction within the previous six months, second or third degree heart block or bundle branch block)
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation; men and women of childbearing potential must be willing to consent to using effective contraception while on treatment and for at least 3 months thereafter; women of childbearing potential must have a negative pregnancy test; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

* All histologies other than squamous cell carcinoma
* Salivary gland and paranasal sinus squamous cell carcinoma
* Patients who have had prior chemotherapy or radiotherapy
* Patients may not be receiving any other investigational agents
* Patients with known brain metastases or direct cerebral invasion by tumor should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events; patients with intracranial extension (but without cerebral involvement) may still be eligible to participate
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to OSI-774 or docetaxel, including other drugs formulated with polysorbate 80
* No pre-existing peripheral neuropathy >= grade 2
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated on this protocol
* HIV positive patients are excluded from participation
* Patients with history of any other malignancy (except squamous cell or basal cell cancer of the skin or CIS of cervix) are ineligible unless a period of 5 years has elapsed since treatment of the previous cancer and the patient has remained continuously disease free
* Patients who are felt to be poorly compliant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2002-09; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
MTD defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity assessed using Common Toxicity Criteria (CTC) version 3.0 (Phase I) | 9 weeks
Pharmacokinetic profile (Phase I) | Pre-dose, 0.5, 1, 2, 4, 8, 12, 24 48, and 72 hours
Time to disease progression (TTP) (Phase II) | Up to 5.5 years

SECONDARY OUTCOMES:
Progression-free survival (PFS) (Phase II) | From the date of treatment to date of death or date of disease progression, and to date of last follow-up for those still alive and progression free, assessed up to 5.5 years
  Will be estimated by Kaplan-Meier method.
Overall survival (OS) (Phase II) | From the date of treatment to date of death, and to date of last follow-up for those still alive, assessed up to 5.5 years
  Will be estimated by Kaplan-Meier method.
True objective response rate (Phase II) | Up to 5.5 years
  Will be estimated based on the number of responses using a binomial distribution and its confidence interval will be estimated using Wilson's method.
Changes of EGFR expression and serum markers over time (Phase II) | Baseline and up to 5.5 years
  The Wilcoxon signed rank test (the non-parametric version of paired T-test) will be used.
Patterns of gene expression data (Phase II) | Up to 5.5 years
  Cluster analysis including hierarchical clustering, Gaussian clustering, k means clustering, will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Panayiotis (Panos) Savvides, Principal Investigator — Case Western Reserve University
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States